CLINICAL TRIAL: NCT02675712
Title: The Effect of African Drumming on on Mental Well-being Among Adults With Acute Mood Disorder
Brief Title: Effect of African Drumming in Mood Disorders
Status: Completed | Type: Observational
Sponsor: University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Dr Nicola Plastow, Lecturer in Occupational Therapy, University of Stellenbosch
Other Study IDs: S15/02/022
Record Dates: First submitted 2016-01-20; First posted 2016-02-05 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Depressive Disorder; Bipolar Disorder
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults with acute mood disorders: Adults aged over 18 diagnosed with an acute episode of a mood disorder using DSM-V criteria
  Interventions: Other: African drumming

INTERVENTIONS:
Other: African drumming — Rhythmic beating or tapping of a variety of percussion instruments, which often occurs within a group setting
  Other Names: Drumming

SUMMARY:
This pilot study evaluated whether participating in an African drumming activity for 45 minutes immediately improved mental well-being among 13 adults diagnosed with acute mood disorders who were attending a private mental health clinic. The drumming intervention was completed by occupational therapists.

DETAILED DESCRIPTION:
This pilot study evaluated the effectiveness of an occupational therapy-led African drumming group on mental well-being among adult psychiatric inpatients with mood disorders. A secondary purpose was to test a protocol for the delivery of African drumming interventions to adults with acute mood disorders.

A quasi-experimental uncontrolled one-group pre-test-post-test design was used to collect data during six drumming groups at an acute mental health clinic. Thirteen adults completed assessments of different aspects of mental well-being, including mood and enjoyment, before and after the intervention. Because this was a pilot study, participants were not assigned to any comparison groups. In addition, in-patients at the clinic received the intervention whether they participated in the study or not.

Improvement in mental well-being across different domains of mental well-being was expected, including feelings of anger, tension, confusion, depression, fatigue and vigour. The researchers also expected the intervention to be more effective in participants with previous drumming experience, and in those with lower levels of anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* Attending mental health clinic
* Diagnosed mood disorder
* Voluntarily attending drumming group

Exclusion Criteria:

* Psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 13 adults diagnosed with a mood disorder (by their own physician), aged 33 to 69 years (M = 45.38, SD = 11.48). The population included both women (n = 10) and men (n = 3). Almost half the participants were of Mixed Ethnicity (n = 6), while the remaining participants were White (n = 7).
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Stellenbosch Mood Scale (STEMS) | Baseline and 45 minutes
  Change from baseline in Stellenbosch Mood Scale at 45 minutes

SECONDARY OUTCOMES:
Generalised Anxiety Disorder - 7 scale (GAD-7) | Baseline
  Level of anxiety as measured by a 7-item self-report Likert-type scale
Primary Health Questionnaire - 9 (PHQ-9) | Baseline
  Level of depression as measured by a 9-item self-report Likert-type scale
Enjoyment of Interaction Scale | 45 minutes
  Enjoyment of the intervention as measured by a 4-item self-report Likert-type scale

CONTACTS AND LOCATIONS:
Overall Officials: Nicola A Plastow, PhD, Principal Investigator — University of Stellenbosch

IPD SHARING:
Plan to Share IPD: No